CLINICAL TRIAL: NCT04535700
Title: Non-blinded, Randomized and Controlled Clinical Trial of Pioglitazone Treatment in Patients With Type 2 Diabetes Mellitus and Covid-19
Brief Title: Clinical Trial of Pioglitazone Treatment in Patients With Type 2 Diabetes Mellitus and Covid-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCORPIO
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes
Keywords: pioglitazone; Covid19
MeSH Terms: conditions — Diabetes Mellitus, Type 2; COVID-19 | interventions — Pioglitazone; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone 30 mg
- Standard of care treatment (Other)
  Interventions: Other: standard of care

INTERVENTIONS:
Drug: Pioglitazone 30 mg — Patients receive 30 mg/day of pioglitazone for the entire period they remain in hospital
  Arms: pioglitazone
Other: standard of care — Patients receive the standard of care, according to the hospital protocol for patients with type 2 diabetes mellitus hospitalized.
  Arms: Standard of care treatment

SUMMARY:
The treatment with pioglitazone added to the standard treatment of patients with DM2 hospitalized for COVID-19 may produce a decrease in the number of patients who progress to a second phase of severe systemic inflammation.

DETAILED DESCRIPTION:
According to the latest studies, the evolution of the SARS-CoV-2 (COVID-19) infection shows two clinically different phases: The first phase of viral and clinical infection of viriasis (fever, myalgia, etc.) affects all patients and it is resolved in asymptomatic patients or with clinically moderate-mild affectations. However, towards the end of the first week of illness, a not inconsiderable number of patients progress towards a second phase of rapid and abrupt deterioration of their respiratory and cardiac function.

More and more data indicate an important role of overactivated macrophages, interleukin 6 (IL6) and an excessive inflammatory response in the genesis of this second phase of aggravation. Linking with this hypothesis, the adipose tissue densely infiltrated by macrophages is the source of one third of the body's IL6, its production being even greater in the fat of central disposition of male distribution. All of this could explain the worse prognosis observed in men, obese and with type 2 diabetes (DM2).

Regarding the possible effect of pioglitazone on the expression of ACE2, there is little literature, and less evidence, about the response of this receptor to treatment with pioglitazone, and what is more important, its effect on COVID-19 infection.

Two studies have analyzed the expression of this receptor after administration of pioglitazone in different murine models of liver and kidney disease. The conclusions of these studies were that the administration of pioglitazone in rats with hepatic steatosis increased the expression of ACE2. It is known that the increased expression of ACE2 facilitates the entry of SARS-CoV-2 into the cell, in animal models it has been seen that ACE2 protects against the development of respiratory distress syndrome and that severe cases of COVID-19 and SARS 2003 have been linked to the possible inhibition of ACE2 by the virus and the increase in angiotensin II.

In conclusion, it is a safe and proven drug in patients with DM2, cheap, with years of clinical experience. The use of pioglitazone added to the conventional treatment of patients at high risk, such as patients with COVID-19 and DM2, could be accompanied by a better evolution of the patients, avoiding or mitigating the inflammatory process that already occurs before its onset. seems to trigger the second accelerated phase of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients > 18 years
2. Confirmed diagnosis of COVID-19 or high clinical suspicion according to current criteria.
3. Diagnosis prior to admission of DM2.
4. Patients who provide their informed consent to participate in the study

Exclusion Criteria:

1. Under 18 years
2. Known hypersensitivity to the active ingredient or any of the drug's excipients.
3. Known history of heart failure or situation at the time of initiation of the heart failure study.
4. Hepatic failure.
5. Dialysis
6. Situation of diabetic ketoacidosis at the start of the study.
7. Diabetes mellitus different from type 2.
8. Active bladder cancer or a history of bladder cancer
9. Hematuria
10. Patients included in another experimental study with another drug.
11. Admission to the Intensive Care Unit.
12. Patients requiring mechanical ventilation at the time of inclusion
13. Pregnancy
14. Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Patients treated with pioglitazone, together with conventional treatment for COVID-19 infection, who during their admission evolve towards the need to receive support with mechanical ventilation, enter the ICU and / or die. | Through hospitalization period, an average of 10-20 days until hospital discharge
  Number of patients receive pioglitazone treatment during their hospital stay who receive support with mechanical ventilation, enter the ICU and / or die.

SECONDARY OUTCOMES:
Incidence of pioglitazone treatment-Emergent Adverse Events in patients with DM2 and symptomatic SARS-CoV-2 infection. | Everyday through hospitalization period, an average of 10-20 days until hospital discharge
  Proportion of patients who develop heart failure or adverse reaction associated with treatment.
Biomarker analysis: systemic inflammation parameters during the administration of pioglitazone treatment. | Each 48 hours through hospitalization period, an average of 10-20 days until hospital discharge
  Changes in this inflammation parameter: C-reactive protein (in mg/dl)
Biomarker analysis: systemic inflammation parameters during the administration of pioglitazone treatment. | Each 48 hours through hospitalization period, an average of 10-20 days until hospital discharge
  Changes in this inflammation parameter: D-dimer (in μg/mL)
Biomarker analysis: systemic inflammation parameters during the administration of pioglitazone treatment. | Each 48 hours through hospitalization period, an average of 10-20 days until hospital discharge
  Changes in this inflammation parameter: ferritin (in ng/mL)
Biomarker analysis: systemic inflammation parameters during the administration of pioglitazone treatment. | Each 48 hours through hospitalization period, an average of 10-20 days until hospital discharge
  Changes in this inflammation parameter: creatine kinase (CK) (in mg/dL)
Biomarker analysis: systemic inflammation parameters during the administration of pioglitazone treatment. | Each 48 hours through hospitalization period, an average of 10-20 days until hospital discharge
  Changes in this inflammation parameter: number of lymphocytes (in μL)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain